CLINICAL TRIAL: NCT01868932
Title: Treating Wheezing in Children With Hypertonic Saline (TWICS)
Acronym: TWICS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding declined. Study never initiated.
Sponsor: Dr. Michael Flavin (Other)
Responsible Party: Sponsor-Investigator, Dr. Michael Flavin, Professor of Pediatrics, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TWICS; HSTWICS (Other: Queen's Department of Pediatrics)
Record Dates: First submitted 2013-05-28; First posted 2013-06-05 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2014-01

CONDITIONS: Wheeze
Keywords: wheeze; early childhood; asthma; bronchiolitis; infection triggered
MeSH Terms: conditions — Respiratory Sounds; Asthma; Bronchiolitis | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypertonic saline (Experimental): inhalation of 4 ml nebulized study solution containing 3% hypertonic saline (HS, study group). Each dose of study solution will also contain a standard dose of bronchodilator (salbutamol, 0.15 mg/kg; 0.03 ml/kg of 0.5% salbutamol nebulizer solution) 1,2 added by the ED staff. Initial therapy will consist of 3 consecutive nebulizations given in rapid succession (back-to-back, approximately every 20 minutes).
  Interventions: Other: hypertonic saline
- saline (Active Comparator): inhalation of 4 ml nebulized study solution containing saline 0.9% saline (NS, control group). Each dose of study solution will also contain a standard dose of bronchodilator (salbutamol, 0.15 mg/kg; 0.03 ml/kg of 0.5% salbutamol nebulizer solution) 1,2 added by the ED staff. Initial therapy will consist of 3 consecutive nebulizations given in rapid succession (back-to-back, approximately every 20 minutes).
  Interventions: Other: saline

INTERVENTIONS:
Other: hypertonic saline — inhaled nebulized 3%NaCl
  Other Names: nebulized hypertonic saline; aerosolized hypertonic saline
  Arms: hypertonic saline
Other: saline — inhaled nebulized 0.9% NaCl
  Other Names: nebulized saline; aerosolized saline
  Arms: saline

SUMMARY:
Hypothesis: substitution of nebulized 3% NaCl (HS) for the standard normal saline (NS) used in bronchodilator therapy for acute viral wheezing in all children under age 6 years will provide superior symptom relief leading to decreased admission rates from the Emergency Department.

The study will test the efficacy of frequent doses of inhaled bronchodilator co-administered with either 3% hypertonic saline (HS, study group) or 0.9% normal saline (NS, control group) in a prospective, double blind, randomized controlled, multi-centre clinical trial of children under age 6 years presenting to the ED with acute viral-associated wheezing.

DETAILED DESCRIPTION:
the brief summary captures the essence of the study

ELIGIBILITY:
Inclusion Criteria:

1. Age under 6 years
2. History of viral upper respiratory infection within previous 7 days
3. Wheezing or crackles detected on chest auscultation
4. Respiratory Distress Assessment Instrument (RDAI) score of 4 or greater or oxygen saturation (SaO2) of 94% or less in room air.

Exclusion Criteria:

1. History of immunodeficiency, chronic cardiopulmonary disease (other than past history of wheezing), Down syndrome, gestational age under 34 weeks.
2. Severe illness at presentation as defined by any of the following

   * respiratory rate greater than 80/min
   * SaO2 less than 88% in room air
   * need for assisted ventilation
3. Use of nebulized HS within previous 12 hours
4. Presence of active varicella infection.

Ages: 2 Days to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Rates of admission to hospital | duration of hospital ER stay, an average of 4 hours
  Rates of admission to hospital

SECONDARY OUTCOMES:
Improvement in respiratory distress scores after initial protocol treatment in the ED | time from pre-intervention assessment to post-intervention assessment, an average of 2 hours
  Improvement in respiratory distress scores after initial protocol treatment in the ED
Length-of-stay in the ED in the subgroup of patients not admitted | an average of 6 hours
  Length-of-stay in the ED in the subgroup of patients not admitted
Cumulative dose of bronchodilator administered in ED prior to admission/discharge order | an average of 6 hours
  Cumulative dose of bronchodilator administered in ED prior to admission/discharge order
Length of hospital stay in the those who are admitted | length of hospital stay, an average of 3 days
  Length of hospital stay in the those who are admitted
Rate of return visit to ED (for respiratory illness) within 14 days of enrollment | 14 days
  Rate of return visit to ED (for respiratory illness) within 14 days of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Flavin, Principal Investigator — Queen's University